CLINICAL TRIAL: NCT04661540
Title: A Single-Blind Dose-Ranging Pharmacodynamic Study of Auxora for the Treatment of Patients With Critical COVID-19 Pneumonia
Brief Title: A Study of Auxora in Patients With Critical COVID-19 Pneumonia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was terminated early due to the limited number of new COVID-19 hospitalizations.
Sponsor: CalciMedica, Inc. (Industry)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: CM4620-205
Record Dates: First submitted 2020-12-04; First posted 2020-12-10 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Pneumonia
Keywords: COVID-19; Coronavirus; Pneumonia; Calcium Release-Activated Calcium Channel (CRAC) Inhibitors; CM4620; Auxora
MeSH Terms: conditions — Pneumonia; COVID-19; Coronavirus Infections | interventions — zegocractin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Auxora (Experimental): Auxora will be given as a continuous infusion:
  Day 1: All 3 cohorts will receive 1.25 mL/kg over 4 hours; After initial infusion is complete, Cohort 3 will receive a continuous infusion of 1.0 mL/kg/24 hours for 96 hours Day 2: Cohort 1 will receive 1.0 mL/kg over 4 hours; Cohort 2 will receive 1.25mL/kg over 4 hours Day 3: Cohort 1 and 2 will receive 1.0 mL/kg over 4 hours Day 4: Cohort 2 will receive 1.0 mL/kg over 4 hours
  Interventions: Drug: CM4620-IE (Injectable Emulsion)
- Placebo (Placebo Comparator): Placebo will be given as a continuous infusion:
  Day 1: All 3 cohorts will receive 1.25 mL/kg over 4 hours. After initial infusion is complete, Cohort 3 will receive a continuous infusion of 1.0 mL/kg/24 hours for 96 hours Day 2: Cohort 1 will receive 1.0 mL/kg over 4 hours; Cohort 2 will receive 1.25mL/kg over 4 hours Day 3: Cohort 1 and 2 will receive 1.0 mL/kg over 4 hours Day 4: Cohort 2 will receive 1.0 mL/kg over 4 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CM4620-IE (Injectable Emulsion) — Auxora is an injectable emulsion containing 1.6mg/ML of the active pharmaceutical ingredient CM4620. Auxora will be administered intravenously as a continuous infusion
  Other Names: Auxora
  Arms: Auxora
Drug: Placebo — Matching placebo is an injectable emulsion containing no active pharmaceutical ingredient. Placebo will be administered intravenously as a continuous infusion
  Arms: Placebo

SUMMARY:
This is a single-blind study of Auxora in patients with critical COVID-19 pneumonia, consisting of up to 3 cohorts of escalating dose. The main goal was to assess pharmacodynamic parameters of immune response, while also assessing safety and tolerability of the drug in this patient population.

DETAILED DESCRIPTION:
The primary objective of this study was to assess the pharmacodynamic response of bronchoalveolar lavage (BAL) T cell/monocyte subsets and chemokine release to various doses of Auxora in patients with critical COVID-19 pneumonia. Other objectives included assessment of safety and tolerability of Auxora in patients with critical COVID-19 pneumonia, as well as pharmacokinetic profile of Auxora in these patients. Efficacy was also to be examined based on all-cause mortality at day 60, number of days on mechanical ventilation after randomization, number of days in the hospital after randomization, and number of days in the ICU after randomization.

Patients were randomized 3:1 to Auxora or Placebo. The first 4 patients were enrolled in Cohort 1 (3 Auxora, 1 Placebo). If dose escalation occurred, the next 4 patients were to be enrolled in Cohort 2. If dose escalation occurred again, the next 8 patients were to be enrolled in Cohort 3. The decision to escalate dosing was made by CalciMedica in consultation with the PI and after the review of safety events in Cohorts 1 and 2.

(Note: Trial terminated early after the first patient was enrolled in Cohort 3 due to lack of new Covid-19 hospitalizations.)

ELIGIBILITY:
Inclusion Criteria:

1. Has laboratory-confirmed SARS-CoV-2 infection as determined by polymerase chain reaction (PCR) or other commercial or public health assay in any specimen;
2. Moderate ARDS characterized by the following criteria:

   * Invasive mechanical ventilation with a minimum PEEP of 5 cm H2O;
   * PaO2/FiO2 ≤200 that may be estimated from pulse oximetry or determined by arterial blood gas;
   * No evidence of volume overload or heart failure;
3. The patient is ≥18 years of age at the time of consent;
4. QTcF interval ≤ 440 milliseconds;
5. A female patient of childbearing potential must not attempt to become pregnant for 39 months, and if sexually active with a male partner, is willing to practice acceptable methods of birth control for 39 months after the last dose of study drug;
6. A male patient who is sexually active with a female partner of childbearing potential is willing to practice acceptable methods of birth control for 39 months after the last dose of study drug. A male patient must not donate sperm for 39 months;
7. The patient is willing and able to, or has a legal authorized representative (LAR) who is willing and able to, provide informed consent to participate, and to cooperate with all aspects of the protocol.

Exclusion Criteria:

1. Expected survival or time to withdrawal of life-sustaining treatments expected to be <7 days.
2. ECMO;
3. Suspected septic shock;
4. The patient has a history of:

   * Organ or hematologic transplant;
   * HIV;
   * Active hepatitis B or hepatitis C infection;
5. Current treatment with:

   * Chemotherapy;
   * Immunosuppressive medications or immunotherapy (see Section 5.3 for list of prohibited immunosuppressive medications and immunotherapy) at the time of consent;
   * Hemodialysis or Peritoneal Dialysis;
6. The patient is known to be pregnant or is nursing;
7. Currently participating in another study of an investigational drug or therapeutic medical device at the time of consent;
8. Allergy to eggs or any of the excipients in study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 10 patients were screened, 1 of which did not meet all inclusion/exclusion criteria, resulting in 9 patients randomized. All 9 completed study treatment, and 0 patients withdrew from the study.
  Patients were randomized 3:1 to Auxora or Placebo. The first 4 patients were enrolled in Cohort 1, and the next 4 in Cohort 2. The next 8 patients were to be enrolled in Cohort 3, but trial terminated early after the first patient was enrolled in Cohort 3, due to lack of new Covid-19 hospitalizations.
Groups:
- Auxora Cohort 1: Auxora will be given as a continuous infusion:
  Day 1: 1.25 mL/kg (2.0 mg/kg) over 4 hours; Day 2: 1.0 mL/kg (1.6 mg/kg) over 4 hours; Day 3: 1.0 mL/kg (1.6 mg/kg) over 4 hours
- Auxora Cohort 2: Auxora will be given as a continuous infusion:
  Day 1: 1.25 mL/kg (2.0 mg/kg) over 4 hours Day 2: 1.25mL/kg (2.0 mg/kg) over 4 hours Day 3: 1.0 mL/kg (1.6 mg/kg) over 4 hours Day 4: 1.0 mL/kg (1.6 mg/kg) over 4 hours
- Auxora Cohort 3: Auxora will be given as a continuous infusion:
  Day 1: Patients will initially receive 1.25 mL/kg (2.0 mg/kg) over 4 hours; After initial infusion is complete, patients will start a continuous infusion of 1.0 mL/kg/24hours for 96 hours (1.6mg/kg/24hours, ending 4 days and 4 hours after the start of first infusion).
- Placebo: Placebo will be given as a continuous infusion, with infusion volume and times matching those of the Auxora Cohort for each respective period.
  Day 1: All patients randomized to placebo will receive 1.25 mL/kg over 4 hours. After initial infusion is complete, patients enrolled during period 3 will then receive a continuous infusion of 1.0 mL/kg/24 hours for 96 hours.
  Day 2: Patients randomized to placebo will receive 1.0 mL/kg over 4 hours if enrolled during Period 1, or 1.25mL/kg over 4 hours if enrolled during Period 2.
  Day 3: Patients randomized to placebo during Periods 1 and 2 will receive 1.0 mL/kg over 4 hours.
  Day 4: Patients randomized to placebo during Period 2 will receive 1.0 mL/kg over 4 hours.
Period: Period 1 (Cohort 1)
Arm/Group | Auxora Cohort 1 | Auxora Cohort 2 | Auxora Cohort 3 | Placebo
Started | 3 | 0 | 0 | 1
Completed | 3 | 0 | 0 | 1
Not Completed | 0 | 0 | 0 | 0
Period: Period 2 (Cohort 2)
Arm/Group | Auxora Cohort 1 | Auxora Cohort 2 | Auxora Cohort 3 | Placebo
Started | 0 | 3 | 0 | 1
Completed | 0 | 3 | 0 | 1
Not Completed | 0 | 0 | 0 | 0
Period: Period 3 (Cohort 3)
Arm/Group | Auxora Cohort 1 | Auxora Cohort 2 | Auxora Cohort 3 | Placebo
Started | 0 (Trial was terminated early after first patient was enrolled in Cohort 3.) | 0 | 1 | 0
Completed | 0 | 0 | 1 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Due to low enrollment trial was terminated early, and Auxora-treated patients from all Cohorts were combined into one arm for analysis. All placebo-treated patients were combined into one control arm as planned.
Groups:
- Auxora Cohort 1: Auxora was given as a continuous infusion:
  Day 1: 1.25 mL/kg (2.0 mg/kg) over 4 hours; Day 2: 1.0 mL/kg (1.6 mg/kg) over 4 hours; Day 3: 1.0 mL/kg (1.6 mg/kg) over 4 hours
- Auxora Cohort 2: Auxora was given as a continuous infusion:
  Day 1: 1.25 mL/kg (2.0 mg/kg) over 4 hours Day 2: 1.25mL/kg (2.0 mg/kg) over 4 hours Day 3: 1.0 mL/kg (1.6 mg/kg) over 4 hours Day 4: 1.0 mL/kg (1.6 mg/kg) over 4 hours
- Auxora Cohort 3: Auxora was given as a continuous infusion:
  Day 1: Patients initially received 1.25 mL/kg (2.0 mg/kg) over 4 hours; After initial infusion is complete, patients started a continuous infusion of 1.0 mL/kg/24hours for 96 hours (1.6mg/kg/24hours, ending 4 days and 4 hours after the start of first infusion).
- Placebo: Placebo was given as a continuous infusion, with infusion volume and times matching those of the Auxora Cohort for each respective period.
  Day 1: All patients randomized to placebo received 1.25 mL/kg over 4 hours. After initial infusion was complete, patients enrolled during period 3 then received a continuous infusion of 1.0 mL/kg/24 hours for 96 hours.
  Day 2: Patients randomized to placebo received 1.0 mL/kg over 4 hours if enrolled during Period 1, or 1.25mL/kg over 4 hours if enrolled during Period 2.
  Day 3: Patients randomized to placebo during Periods 1 and 2 received 1.0 mL/kg over 4 hours.
  Day 4: Patients randomized to placebo during Period 2 received 1.0 mL/kg over 4 hours.
- Total: Total of all reporting groups
Arm/Group | Auxora Cohort 1 | Auxora Cohort 2 | Auxora Cohort 3 | Placebo | Total
Number analyzed (Participants) | 3 | 3 | 1 | 2 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (5.2) | 67.0 (3.0) | 46 (NA) — Standard deviation cannot be calculated based on 1 data point. | 54 (1.4) | 57 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 1 | 3
  Male | 2 | 2 | 1 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 1 | 0 | 6
  Not Hispanic or Latino | 1 | 0 | 0 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 1 | 2 | 0 | 1 | 4
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 1 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 1 | 2 | 9
Height [Mean (Standard Deviation); unit: cm] | 170.3 (16.6) | 164.7 (5.8) | 183 (NA) — Standard deviation cannot be calculated based on 1 data point. | 184.0 (12.7) | 172.9 (13.0)
Weight [Mean (Standard Deviation); unit: kg] | 96.7 (26.5) | 78.0 (4.4) | 163.4 (NA) — Standard deviation cannot be calculated based on 1 data point. | 103.5 (26.2) | 99.4 (30.9)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 33.2 (6.6) | 28.9 (1.6) | 48.9 (NA) — Standard deviation cannot be calculated based on 1 data point. | 30.3 (3.6) | 32.9 (7.3)
Number of Participants with Additional Prior Positive Covid Test [Count of Participants; unit: Participants]
  Yes | 3 | 3 | 0 | 1 | 7
  Unknown | 0 | 0 | 0 | 1 | 1
  No | 0 | 0 | 1 | 0 | 1
Number of Participants with Upper Respiratory Co-detection of Sars-CoV-2 [Count of Participants; unit: Participants] | 0 | 1 | 0 | 2 | 3
Number of Participants with Bacterial Superinfection at Intubation [Count of Participants; unit: Participants] | 1 | 1 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Combined CD4, CD8, and Monocyte Cell Population in BAL Fluid, as a Percent of Total WBC Population.
Description: Pharmacodynamic endpoint: Assessment of pharmacodynamic response of bronchoalveolar lavage (BAL) T cell/monocyte subsets to Auxora treatment. Flow cytometry was performed on fluid collected from the BAL performed prior to the SFISD (-12 hours) and 24 (±12) hours after completing the last infusion of study drug in Cohorts 1 and 2 and during the final 24 hours of the continuous infusion in Cohort 3. The percentage of total WBC population was assessed for the combined CD4, CD8, and monocyte cell population, and the change between Pre- and Post-Infusion samples (Post value minus Pre value) was reported.
Time Frame: Baseline Assessment up to 120 hours
Measure: Mean (Standard Deviation); unit: Percent of total WBC population
Arm/Group | Auxora Cohort 1 | Auxora Cohort 2 | Auxora Cohort 3 | Placebo
Number analyzed (Participants) | 3 | 3 | 1 | 2
Percent of total WBC population | -5.6 (31.6) | -7.2 (10.7) | 27.1 (NA) — Standard deviation cannot be calculated from 1 data point. | 22.8 (9.7)

2. Secondary Outcome: Change From Baseline in Percent of Immune Cells in BAL Fluid
Description: Pharmacodynamic endpoint: Assessment of pharmacodynamic response of bronchoalveolar lavage (BAL) T cell/monocyte subsets to Auxora treatment. Flow cytometry was performed on fluid collected from the BAL performed prior to the SFISD (-12 hours) and 24 (±12) hours after completing the last infusion of study drug in Cohorts 1 and 2 and during the final 24 hours of the continuous infusion in Cohort 3. The percentage of total WBC population was assessed for immune cell types and the change between Pre- and Post-Infusion samples (Post value minus Pre value) was reported.
Time Frame: Baseline Assessment up to 120 hours
Measure: Mean (Standard Deviation); unit: Percent of total WBC population
Arm/Group | Auxora Cohort 1 | Auxora Cohort 2 | Auxora Cohort 3 | Placebo
Number analyzed (Participants) | 3 | 3 | 1 | 2
Percent of total WBC population
  CD4 T Cells | -2.4 (15.7) | -3.4 (6.3) | 5.9 (NA) — Standard deviation cannot be calculated from a single data point. | 17.9 (5.4)
  CD8 T Cells | -2.0 (12.5) | -0.5 (4.6) | 23.1 (NA) — Standard deviation cannot be calculated from a single data point. | 5.3 (3.9)
  Neutrophils | -14.5 (43.9) | 24.4 (47.1) | -4.2 (NA) — Standard deviation cannot be calculated from a single data point. | -25.7 (24.0)
  NK cells | -0.2 (1.5) | -1.8 (1.5) | 0.1 (NA) — Standard deviation cannot be calculated from a single data point. | 0.3 (1.3)
  Monocytes | -1.2 (10.0) | -3.3 (5.8) | -13.4 (NA) — Standard deviation cannot be calculated from a single data point. | -0.4 (0.3)
  B cells | 14.2 (10.4) | -12.4 (14.3) | 3.2 (NA) — Standard deviation cannot be calculated from a single data point. | -23.2 (29.9)
  Macrophages | 6.3 (20.0) | -2.3 (23.1) | -3.8 (NA) — Standard deviation cannot be calculated from a single data point. | 25.2 (16.9)

3. Secondary Outcome: Number of Patients Alive at Day 60
Description: Efficacy endpoint: All-cause Mortality at Day 60
Time Frame: Randomization through Day 60
Measure: Count of Participants; unit: Participants
Groups:
- Auxora (ALL): Combined Total data for Auxora-treated patients from all 3 Cohorts.
Arm/Group | Auxora (ALL) | Auxora Cohort 1 | Auxora Cohort 2 | Auxora Cohort 3 | Placebo
Number analyzed (Participants) | 7 | 3 | 3 | 1 | 2
Participants | 3 | 1 | 1 | 1 | 1

4. Secondary Outcome: Number of Days Alive and Out of the Intensive Care Unit (ICU)
Description: Efficacy Endpoint: Days in ICU (after randomization)
Time Frame: From randomization until discharge from ICU, assessed up to 60 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Auxora (ALL) | Auxora Cohort 1 | Auxora Cohort 2 | Auxora Cohort 3 | Placebo
Number analyzed (Participants) | 7 | 3 | 3 | 1 | 2
days | 4.6 (8.0) | 6.3 (11.0) | 0 (0) | 13.0 (NA) — Standard deviation cannot be calculated off of 1 data point. | 0 (0)

5. Secondary Outcome: Number of Days Alive and Out of the Hospital
Description: Efficacy endpoint: Days hospitalized (after randomization)
Time Frame: From randomization until discharge from the hospital, assessed up to 60 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Auxora (ALL) | Auxora Cohort 1 | Auxora Cohort 2 | Auxora Cohort 3 | Placebo
Number analyzed (Participants) | 7 | 3 | 3 | 1 | 2
days | 1.0 (2.6) | 0 (0) | 0 (0) | 7.0 (NA) — Standard deviation cannot be calculated off of 1 data point. | 0 (0)

6. Secondary Outcome: Number of Days Alive and Off Mechanical Ventilation
Description: Efficacy endpoint: Ventilator-free days (after randomization)
Time Frame: From randomization until patient is extubated, assessed up to 60 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Auxora (ALL) | Auxora Cohort 1 | Auxora Cohort 2 | Auxora Cohort 3 | Placebo
Number analyzed (Participants) | 7 | 3 | 3 | 1 | 2
days | 5.9 (10.2) | 8.0 (13.9) | 0 (0) | 17.0 (NA) — Standard deviation cannot be calculated off of 1 data point. | 0 (0)

7. Other Pre Specified Outcome: Number of Patients Experiencing an AE Considered Possibly Related to Study Drug
Description: Safety endpoint. Examines the relatedness of AEs to study drug by assessing the number of patients experiencing any AE (serious or non-serious) considered possibly related to Study Drug.
Time Frame: Randomization through Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Auxora (ALL) | Auxora Cohort 1 | Auxora Cohort 2 | Auxora Cohort 3 | Placebo
Number analyzed (Participants) | 7 | 3 | 3 | 1 | 2
Participants
  Possibly related SAEs | 0 | 0 | 0 | 0 | 0
  Possibly related non-serious AEs | 2 | 1 | 0 | 1 | 0

8. Other Pre Specified Outcome: Number of Patients Experiencing an SAE (at Least 1)
Description: Safety Endpoint: Incidence of treatment emergent Serious Adverse Events (SAEs)
Time Frame: Randomization through day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Auxora (ALL) | Auxora Cohort 1 | Auxora Cohort 2 | Auxora Cohort 3 | Placebo
Number analyzed (Participants) | 7 | 3 | 3 | 1 | 2
Participants | 4 | 1 | 3 | 0 | 2

9. Other Pre Specified Outcome: Intensity of AEs
Description: Safety endpoint: Count of the number of AEs for each level of intensity: mild, moderate, or severe
Time Frame: Randomization through Day 30
Measure: Number; unit: Adverse Events
Arm/Group | Auxora (ALL) | Auxora Cohort 1 | Auxora Cohort 2 | Auxora Cohort 3 | Placebo
Number analyzed (Participants) | 7 | 3 | 3 | 1 | 2
Adverse Events
  Mild | 13 | 2 | 9 | 2 | 5
  Moderate | 21 | 11 | 8 | 2 | 7
  Severe | 8 | 2 | 6 | 0 | 2

10. Other Pre Specified Outcome: Number of Patients Experiencing Pre-defined Changes in Cardiac Conduction Assessed by ECG
Description: Safety endpoint: Patients experiencing Changes in cardiac conduction, defined as: QTcF interval of ≥ 500 msec; QTcF prolongation of ≥ 60 msec as compared to baseline; Mobitz Type II second degree atrioventricular (AV) block; Third degree or high grade AV block; or Polymorphic Ventricular Tachycardia
Time Frame: From randomization up to 144 hours after SFISD (start of first infusion of study drug)
Measure: Count of Participants; unit: Participants
Arm/Group | Auxora (ALL) | Auxora Cohort 1 | Auxora Cohort 2 | Auxora Cohort 3 | Placebo
Number analyzed (Participants) | 7 | 3 | 3 | 1 | 2
Participants | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from randomization through Day 30. All-Cause Mortality was assessed from randomization through Day 60.
Description: Per the protocol, adverse events were assessed from randomization through Day 30 only. An additional mortality assessment was performed at Day 60 for efficacy purposes only. (Note: 3 deaths had occurred in the Auxora-treated group and 1 death in the placebo group by Day 30. 1 additional death had occurred in the Auxora-treated group at the Day 60 mortality assessment.)
Arm/Group | Auxora (ALL) | Auxora Cohort 1 | Auxora Cohort 2 | Auxora Cohort 3 | Placebo
All-Cause Mortality (participants affected / at risk) | 4/7 | 2/3 | 2/3 | 0/1 | 1/2
Serious Adverse Events (participants affected / at risk) | 4/7 | 1/3 | 3/3 | 0/1 | 2/2
Other Adverse Events (participants affected / at risk) | 7/7 | 3/3 | 3/3 | 1/1 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Auxora (ALL) (N=7) | Auxora Cohort 1 (N=3) | Auxora Cohort 2 (N=3) | Auxora Cohort 3 (N=1) | Placebo (N=2)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Distributive shock (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Auxora (ALL) (N=7) | Auxora Cohort 1 (N=3) | Auxora Cohort 2 (N=3) | Auxora Cohort 3 (N=1) | Placebo (N=2)
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 (0) | 1 (1) | 0 (0) | 0
Hypertransaminasemia (Hepatobiliary disorders) | 4 | 2 | 1 | 1 | 1
Systemic candida (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Enterococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Staphylococcal bacteremia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 0 | 0 | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0
Cystitis escherichia (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0
Bronchopulmonary aspergillosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Enterobacter pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 3 | 0 | 0
Lung abscess (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 2 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Pneumonia pseudomonal (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Pneumonia staphylococcal (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1 | 1
Pneumonia streptococcal (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 1
Venous thrombosis (Vascular disorders) | 3 | 1 | 2 | 0 | 1
Superficial vein thrombosis (Vascular disorders) | 1 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
This trial was terminated early due to the limited number of new COVID-19 hospitalizations, leading to small numbers of subjects analyzed (7 randomized to Auxora and 2 randomized to placebo). Hence, no formal hypothesis testing was performed. All performed analyses were based on descriptive summaries.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI shall submit copies of the proposed results communications to the Sponsor at least 30 days in advance of the submission of any proposed publication to a journal, editor, or other third party. Sponsor may request that Confidential Information (other than Study Data) be removed from communications, or that the PI refrain from publication for an additional 60 days in order for patent application(s) directed to the patentable subject matter to be filed with the appropriate patent office(s).

DOCUMENTS (3):
  • Study Protocol (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/40/NCT04661540/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/40/NCT04661540/SAP_001.pdf
  • Informed Consent Form (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/40/NCT04661540/ICF_002.pdf